CLINICAL TRIAL: NCT02469233
Title: A Transdiagnostic Sleep and Circadian Treatment to Improve Community SMI Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Alameda County Behavioral Health Care Services (Unknown); University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH105513 (NIH)
Record Dates: First submitted 2015-06-09; First posted 2015-06-11 (Estimated); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders | interventions — Sleep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TranS-C (Experimental): The Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) is comprised of cross-cutting interventions, 'core modules' and 'optional modules'. TranS-C is derived and adapted from our previous disorder-focused research, firmly grounded in basic science and treatment literature.
  Interventions: Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction
- UC-DT (Active Comparator): Usual Care, Delayed Treatment (DT) is comprised of a case manager who co-ordinates care and refers each client for a medication review and to rehabilitation programs. At the end of 6-months in UC-DT, the participants will receive TranS-C.
  Interventions: Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction

INTERVENTIONS:
Behavioral: Transdiagnostic Intervention for Sleep and Circadian Dysfunction — The intervention is a modular treatment composed of core modules that are given to all participants and modules that are delivered based on the need/s of the participants. The interventions are all cognitive behavioral.

SUMMARY:
Mental illness is often severe, chronic and difficult to treat. The sleep disturbance commonly experienced by individuals with a severe mental illness reduces capacity to function and contributes to key symptoms. This study seeks to determine if an intervention to improve sleep can improve functioning and reduce symptoms and impairment. The investigators will conduct this study in community mental health centers to ensure that the results contribute to closing the worrisome gap between research and practice and to ensure that the findings are generalizable to the real world.

DETAILED DESCRIPTION:
Despite advances in treatment, severe mental illness (SMI) remains common, chronic and difficult to treat. SMI is defined as having at least one mental disorder that lasts for 12-months and leads to substantial life interference. Sleep and circadian dysfunctions are among the most prominent correlates of SMI, yet have been minimally studied in ways that reflect the complexity of the sleep problems experienced by people with SMI. In SMI, sleep and circadian dysfunction undermines affect regulation, cognitive function and physical health, predicts onset and worsening of symptoms and is often chronic even with evidence-based SMI treatment. Prior treatment studies have been disorder-focused-they have treated a specific sleep problem (e.g., insomnia) in a specific diagnostic group (e.g., depression). However, real life sleep and circadian problems are not so neatly categorized, particularly in SMI where features of insomnia overlap with hypersomnia, delayed sleep phase and irregular sleep-wake schedules. Accordingly, the investigators aim to test the hypothesis that a Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) will improve functional impairment, disorder-focused symptoms and sleep and circadian functioning. The investigators will recruit participants across Diagnostic and Statistical Manual of Mental Disorders (DSM) diagnoses and across common sleep and circadian problems. The elements of TranS-C are efficacious across SMI in research settings with research-based providers. The next step is to test TranS-C in community settings with community-based providers. Accordingly, the investigators propose to conduct an 'efficacy in the real world' randomized controlled trial within Alameda County Behavioral Health Care Services (ACBHCS), the community mental health center (CMHC) for Alameda County. The investigators will recruit 120 adults diagnosed with SMI and sleep and circadian dysfunction within ACBHCS. Individuals will be randomly allocated to TranS-C (n = 60) or 6-months of Usual Care followed by Delayed Treatment with TranS-C (UC-DT; n = 60). TranS-C is modularized and delivered across eight to twelve 50-minute, weekly, individual sessions. All participants will be assessed before, immediately following treatment (ie. 9-14 weeks later) and again 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* English language fluency
* Presence of at least one DSM-V mental disorder for 12 months
* One or more of the following sleep or circadian problems for 3 month as assessed with the Sleep and Circadian Problems Interview:

  * ≥30 mins to get to sleep , 3 or more nights per week
  * Waking in the middle of the night for ≥30 minutes, 3 or more nights per week
  * Obtaining less than 6 hours of sleep per night, 3 or more nights per week
  * Obtaining more than 9 hours of sleep per 24 hour period (i.e., nighttime sleep plus daytime napping), 3 or more nights per week
  * More than 2.78 hours of variability in sleep-wake schedule across one week
  * Bedtime later than 2 am, 3 or more nights per week
* Guaranteed bed to sleep in for the duration of the treatment phase
* Receiving care for SMI at ACBHCS and consent to regular communications between research team and psychiatrist and/or case manager

Exclusion Criteria:

* Presence of an active and progressive physical illness or neurological degenerative disease AND/OR substance abuse/dependence making participation in the study unfeasible.
* Current serious suicide risk (assessed by our staff, a case manager or psychiatrist) or homicide risk (assessed by our staff, a case manager or psychiatrist)
* Night shift work >2 nights per week in the past 3 months
* Pregnancy or breast-feeding
* Not able/willing to participate in and/or complete the pre-treatment assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2019-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison G Harvey, PhD, Principal Investigator — University of California, Berkeley
Locations (1):
- Alameda Country Behavioral Health Care Services, Oakland, California, United States

REFERENCES:
- [Derived] Callaway CA, Sarfan LD, Gumport NB, Harvey AG. The impact of module dosage on treatment response in a modular transdiagnostic intervention for sleep and circadian dysfunction (TranS-C). Behav Res Ther. 2023 Sep;168:104368. doi: 10.1016/j.brat.2023.104368. Epub 2023 Jul 5. PMID 37478529
- [Derived] Harvey AG, Dong L, Hein K, Yu SH, Martinez AJ, Gumport NB, Smith FL, Chapman A, Lisman M, Mirzadegan IA, Mullin AC, Fine E, Dolsen EA, Gasperetti CE, Bukosky J, Alvarado-Martinez CG, Kilbourne AM, Rabe-Hesketh S, Buysse DJ. A randomized controlled trial of the Transdiagnostic Intervention for Sleep and Circadian Dysfunction (TranS-C) to improve serious mental illness outcomes in a community setting. J Consult Clin Psychol. 2021 Jun;89(6):537-550. doi: 10.1037/ccp0000650. PMID 34264701
- [Derived] Gumport NB, Yu SH, Harvey AG. Implementing a transdiagnostic sleep and circadian intervention in a community mental health setting: A qualitative process evaluation with community stakeholders. Psychiatry Res. 2020 Nov;293:113443. doi: 10.1016/j.psychres.2020.113443. Epub 2020 Aug 31. PMID 32890862
- [Derived] Harvey AG, Hein K, Dong L, Smith FL, Lisman M, Yu S, Rabe-Hesketh S, Buysse DJ. A transdiagnostic sleep and circadian treatment to improve severe mental illness outcomes in a community setting: study protocol for a randomized controlled trial. Trials. 2016 Dec 20;17(1):606. doi: 10.1186/s13063-016-1690-9. PMID 27998295

RESULTS

PARTICIPANT FLOW:
Groups:
- TranS-C: The 'Transdiagnostic' Intervention for Sleep and Circadian Dysfunction (TranS-C) is comprised of cross-cutting interventions, 'core modules' and 'optional modules'. TranS-C is derived and adapted from our previous disorder-focused research, firmly grounded in basic science and treatment literature.
  Transdiagnostic Intervention for Sleep and Circadian Dysfunction: The intervention is a modular treatment composed of core modules that are given to all participants and modules that are delivered based on the need/s of the participants. The interventions are all cognitive behavioral.
Period: Overall Study
Arm/Group | TranS-C | UC-DT
Started | 61 | 60
Received Allocated Intervention | 59 | 60
Completed Post-assessment | 49 | 58
Completed Follow-up | 53 | 57
Analyzed | 61 | 60
Completed (Completed 6-month follow-up) | 53 | 57
Not Completed | 8 | 3
Not completed — Death | 1 | 1
Not completed — Lost to post or 6 month follow up | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- UC-DT: Usual Care, Delayed Treatment (UC-DT) is comprised of a case manager who co-ordinates care and refers each client for a medication review and to rehabilitation programs. At the end of 6-months in UC-DT, the participants will receive TranS-C.
  Transdiagnostic Intervention for Sleep and Circadian Dysfunction: The intervention is a modular treatment composed of core modules that are given to all participants and modules that are delivered based on the need/s of the participants. The interventions are all cognitive behavioral.
- Total: Total of all reporting groups
Arm/Group | UC-DT | TranS-C | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.45 (13.25) | 47.97 (11.51) | 46.72 (12.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 30 | 63
  Male | 27 | 31 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 51 | 50 | 101
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 4 | 8
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 3
  Black or African American | 26 | 26 | 52
  White | 21 | 25 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 61 | 121
Civil status [Count of Participants; unit: Participants]
  Single | 42 | 38 | 80
  Married/common law partner | 4 | 5 | 9
  Separated/divorced/widowed | 14 | 18 | 32
Education [Count of Participants; unit: Participants]
  High school or below | 22 | 19 | 41
  Vocational school | 2 | 9 | 11
  Some college or completed college | 34 | 30 | 64
  Graduate school | 2 | 3 | 5
Employment [Count of Participants; unit: Participants]
  Full-time | 1 | 1 | 2
  Part-time | 6 | 9 | 15
  Unemployed | 49 | 49 | 98
  Other | 4 | 1 | 5
  Missing | 0 | 1 | 1
Living arrangement [Count of Participants; unit: Participants] — Note: Supported housing includes living in board & care homes, senior housing, transitional housing, and homeless shelters.
  Participants
    Alone | 12 | 8 | 20
    With family (spouse or children) | 8 | 6 | 14
    With friend or roommate or pet | 11 | 11 | 22
    Supported housing | 29 | 35 | 64
    Missing | 0 | 1 | 1
MINI Diagnosis at pre-treatment (current or past) [Count of Participants; unit: Participants] — The Mini-International Neuropsychiatric Interview (MINI; DSM-5, Version 7.0.0 including Schizophrenia and Psychotic Disorders) was included as an evaluation of the presence of current and past Severe mental illness. Note: Comorbidity was common
  Participants
    Schizophrenia spectrum disorder | 29 | 26 | 55
    Bipolar disorder | 13 | 21 | 34
    Major depressive disorder | 17 | 11 | 28
    Any anxiety disorder | 27 | 30 | 57
    Obsessive compulsive disorder | 12 | 9 | 21
    Post-traumatic stress disorder | 12 | 6 | 18
    Substance use disorder | 20 | 19 | 39
    Psychotic symptoms/features | 42 | 39 | 81
DUKE diagnoses at pre-treatment (current) [Count of Participants; unit: Participants] — Duke Structured Interview for Sleep Disorders (DUKE) diagnoses at pre-treatment (current): The diagnostic measure for sleep disorders was the Duke Structured Interview for Sleep Disorders. Note: Comorbidity was common
  Participants
    Insomnia disorder | 49 | 52 | 101
    Hypersomnolence disorder | 14 | 17 | 31
    Circadian Rhythm Disorder: Delayed sleep phase type | 5 | 3 | 8
    Circadian Rhythm Disorder: Advanced sleep phase type | 0 | 2 | 2
    Circadian Rhythm Disorder: Irregular sleep-wake type | 0 | 1 | 1
    Circadian Rhythm Disorder: Restless leg syndrome | 3 | 2 | 5
    Circadian Rhythm Disorder: Periodic limb movement disorder | 4 | 1 | 5
Education (in years) [Mean (Standard Deviation); unit: Years] | 13.38 (3.89) | 13.80 (3.05) | 13.59 (3.48)
Annual personal income [Mean (Standard Deviation); unit: Dollars ($)] | 12,429 (15,317) | 12,636 (9,850) | 12,531 (12,838)
Annual household income [Mean (Standard Deviation); unit: Dollars ($)] | 24,091 (27,507) | 26,537 (23,576) | 25,216 (25,546)

OUTCOME MEASURES:

1. Primary Outcome: Impairment (Sheehan Disability Scale)
Description: Sheehan Disability Scale (SDS) (sleep). 3-item. The SDS evaluates the extent to which work/school, social life, and home/ family responsibilities are impaired on a 0-10 (not at all to extremely) scale. The 3-items are summed to compute the total score and assess global functional impairment. Scores can range from 0 to 30, with higher values indicating higher impairment.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: Although all randomized participants were included in the intent-to-treat analysis, the "Number Analyzed" represents participants who contributed data at each time point. Differences from the overall number analyzed reflect missing assessments due to attrition.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
score on a scale
  Pre treatment | 14.30 (8.51) | 12.03 (6.20)
  Post treatment: number analyzed (Participants) | 58 | 49
  Post treatment | 11.76 (7.57) | 6.57 (7.07)
  6-month follow-up: number analyzed (Participants) | 57 | 53
  6-month follow-up | 10.51 (8.36) | 7.00 (6.41)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.025, Intent-to-treat, multilevel modeling; Using intent-to-treat, multilevel modeling with maximum likelihood estimation with the assumption of missing at random, to examine continuous outcomes; Time by treatment interaction coeff. = -3.18
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.28, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -1.52

2. Primary Outcome: Disorder-Focused Composite Score (DSM-5)
Description: DSM-5 Cross Cutting Measure. 23-items. Individuals report how much each domain has bothered them in the last 2 weeks on a 0-4 scale (not at all to nearly every day). The total score is calculated by summing the highest score in each of the 13 domains (depression, anger, mania, anxiety, somatic symptoms, suicidal ideation, psychosis, sleep problems, memory, repetitive thoughts and behaviors, dissociation, personality functioning, and substance use). Total scores can range from 0 to 52, with higher scores indicating greater severity of impairment. is rated on a 5-point scale, with higher scores indicating more severe impairment.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
score on a scale
  Pre treatment | 25.57 (10.72) | 25.05 (9.75)
  Post treatment: number analyzed (Participants) | 58 | 49
  Post treatment | 23.53 (10.59) | 17.00 (11.23)
  6-month follow-up: number analyzed (Participants) | 57 | 53
  6-month follow-up | 23.07 (9.78) | 18.67 (11.38)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.001, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; time by treatment interaction coeff. = -5.88
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.03, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; maximum likelihood estimation = -3.90

3. Primary Outcome: Sleep and Circadian Function: PROMIS-Sleep Disturbance
Description: PROMIS-Sleep Disturbance (PROMIS = Patient-Reported Outcomes Measurement Information System). The 8-item short version assesses sleep disturbance over the past 7 days, including restlessness, sleep quality, ability to fall and stay asleep, and refreshment following sleep using a 1-5 scale (not at all or never to very much or always). Scores range from 8 to 40, with higher scores indicating increased disturbance.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
score on a scale
  PROMIS-Sleep Disturbance (Pre) | 29.02 (6.57) | 28.26 (6.06)
  PROMIS-Sleep Disturbance (Post): number analyzed (Participants) | 58 | 49
  PROMIS-Sleep Disturbance (Post) | 27.33 (7.22) | 20.88 (8.91)
  PROMIS-Sleep Disturbance (6-month follow-up): number analyzed (Participants) | 57 | 53
  PROMIS-Sleep Disturbance (6-month follow-up) | 26.40 (8.00) | 20.87 (8.50)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p < 0.0001, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; time by treatment interaction coeff. = -5.55
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p < 0.0001, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -4.92

4. Primary Outcome: Sleep and Circadian Function: PROMIS-Sleep-Related Impairment
Description: PROMIS-Sleep-Related Impairment (PROMIS = Patient-Reported Outcomes Measurement Information System). 16-item. Scores range from 16 to 80, with higher scores indicating increased disturbance.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
score on a scale
  PROMIS-Sleep-Related Impairment (Pre) | 51.02 (14.09) | 47.93 (11.80)
  PROMIS-Sleep-Related Impairment (Post): number analyzed (Participants) | 58 | 49
  PROMIS-Sleep-Related Impairment (Post) | 47.22 (14.14) | 35.16 (14.01)
  PROMIS-Sleep-Related Impairment (6-month follow-up): number analyzed (Participants) | 57 | 53
  PROMIS-Sleep-Related Impairment (6-month follow-up) | 44.30 (15.22) | 35.65 (13.83)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p < 0.0001, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -9.14
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.027, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -5.37

5. Secondary Outcome: Depression (QIDS)
Description: QIDS (Quick Inventory of Depressive Symptoms). 16-item instrument assessing depressive symptoms. Each item is rated on a 4-point scale (0-3), with higher scores indicating greater symptom severity.
  Scoring involves summing the highest score from each of the 9 DSM-IV Major Depressive Disorder symptom domains (sleep, weight, psychomotor changes, depressed mood, decreased interest, fatigue, guilt, concentration, and suicidal ideation). Total scores range from 0 (Normal/No Depression) to 27 (Very Severe Depression). Higher scores indicate greater severity of depressive symptoms.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
score on a scale
  Pre-treatment | 12.50 (4.71) | 12.03 (5.15)
  Post-treatment: number analyzed (Participants) | 58 | 49
  Post-treatment | 10.55 (5.54) | 8.88 (5.70)
  6-month follow-up: number analyzed (Participants) | 57 | 53
  6-month follow-up | 10.67 (4.58) | 8.46 (5.03)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.32, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.95
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.08, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -1.67

6. Secondary Outcome: Substance Use (ASSIST )
Description: ASSIST (Alcohol, Smoking and Substance Involvement Screening Test). Frequency of use, substance dependence, and related health, social, legal, financial, and employment problems in the past 3 months are rated on a 5-point scale (never to daily of almost daily). Problems with family and friends caused by substance use and failed attempts to cut down or quit substance use are measured on a 3-point scale (no, never, yes, in the past 3 months, yes, but not in the past 3 months). The total risk score is calculated by summing scores across all drug categories, with total scores ranging from 0 to 414. Higher scores indicate greater substance-related risks and problems.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
score on a scale
  Pre-treatment | 33.68 (25.87) | 39.70 (26.68)
  Post-treatment: number analyzed (Participants) | 58 | 49
  Post-treatment | 14.62 (17.15) | 15.35 (17.13)
  6-month follow-up: number analyzed (Participants) | 57 | 53
  6-month follow-up | 32.58 (25.25) | 34.60 (24.10)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.72, intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.09
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.74, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.08

7. Secondary Outcome: Psychotic Symptoms (PSYRATS )
Description: PSYRATS (Psychotic Symptom Rating Scales). Each of the 17 items is rated on a 5-point scale from 0 (absent) to 4 (severe). Scores are summed for auditory hallucinations (sum of 11 items) and delusions (sum of 6 items). Total scores range from 0 to 68, with higher scores indicating greater severity of psychotic symptoms.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
score on a scale
  Pre-treatment | 36.60 (5.13) | 39.60 (14.29)
  Post-treatment: number analyzed (Participants) | 58 | 49
  Post-treatment | 41.73 (11.39) | 36.00 (14.82)
  6-month follow-up: number analyzed (Participants) | 57 | 53
  6-month follow-up | 42.58 (9.44) | 25.80 (11.23)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.73, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -2.46
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.02, intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -17.52

8. Secondary Outcome: Means and Variability of Sleep Efficiency (Daily Sleep Diary)
Description: Sleep efficiency (SE), calculated as total sleep time divided by time in bed, multiplied by 100, was recorded via sleep diary over 7 consecutive days. For each participant, the mean and within-person standard deviation (SD) of SE were calculated across the days to reflect an average and night-to-night variability. Group-level outcomes reflect the average of these participant-level means and SDs.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of sleep efficiency
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
percentage of sleep efficiency
  SE mean at Pre-treatment | 77.61 (11.89) | 77.39 (13.52)
  SE variability at Pre-treatment | 12.52 (7.63) | 11.92 (6.71)
  SE mean at Post-treatment: number analyzed (Participants) | 58 | 49
  SE mean at Post-treatment | 78.93 (14.50) | 84.31 (10.07)
  SE variability at Post-treatment: number analyzed (Participants) | 58 | 49
  SE variability at Post-treatment | 11.86 (8.49) | 10.01 (7.95)
  SE mean at 6-month follow-up: number analyzed (Participants) | 57 | 53
  SE mean at 6-month follow-up | 79.54 (12.88) | 84.78 (10.86)
  SE variability at 6-month follow-up: number analyzed (Participants) | 57 | 53
  SE variability at 6-month follow-up | 11.25 (6.71) | 9.24 (7.87)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; SE mean (min): Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.03, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = 5.68
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; SE mean (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.03, intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = 5.89
Statistical Analysis 3: Comparison: UC-DT vs TranS-C; SE variability (min): Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.43, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -1.45
Statistical Analysis 4: Comparison: UC-DT vs TranS-C; SE variability (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.40, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -1.55

9. Secondary Outcome: Actigraphy Measured Sleep (TST)
Description: Actigraphy-derived total sleep time (TST) is the total amount of sleep obtained by the participant per 24 hrs, which was recorded daily over a 1-week period per timepoint. For each participant, the mean and standard deviation (SD) of TST were calculated across the days. Group-level outcomes reflect the average of these participant-level means and SDs.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
Minutes
  TST mean at Pre-treatment | 421.35 (126.92) | 453.65 (147.28)
  TST variability at Pre-treatment | 132.08 (75.83) | 132.34 (79.71)
  TST mean at Post-treatment: number analyzed (Participants) | 58 | 49
  TST mean at Post-treatment | 411.82 (108.28) | 427.23 (135.85)
  TST variability at Post-treatment: number analyzed (Participants) | 58 | 49
  TST variability at Post-treatment | 135.38 (75.05) | 140.06 (95.02)
  TST mean at 6-month follow-up: number analyzed (Participants) | 57 | 53
  TST mean at 6-month follow-up | 443.24 (119.47) | 437.69 (137.88)
  TST variability at 6-month follow-up: number analyzed (Participants) | 57 | 53
  TST variability at 6-month follow-up | 144.86 (88.72) | 134.43 (96.75)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; TST mean (min): Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.59, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -12.68
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; TST mean (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.22, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -28.33
Statistical Analysis 3: Comparison: UC-DT vs TranS-C; TST variability (min) : Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.80, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = 4.65
Statistical Analysis 4: Comparison: UC-DT vs TranS-C; TST variability (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.68, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -7.57

10. Secondary Outcome: Daytime Activity (Actigraphy)
Description: Daytime activity was measured via actigraphy over 7 consecutive days per timepoint. For each participant, their daily waking activity counts were extracted, and the mean and within-person standard deviation (SD) of these counts were calculated across 7 days. Group-level outcomes reflect the average of these participant-level means and SDs.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Activity counts
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
Activity counts
  Count Mean at Pre-treatment | 1309.74 (532.79) | 1280.09 (607.46)
  Count Variability at Pre-treatment | 379.69 (211.65) | 394.04 (256.07)
  Count Mean at Post-treatment: number analyzed (Participants) | 58 | 49
  Count Mean at Post-treatment | 1361.19 (532.36) | 1257.82 (680.06)
  Count Variability at Post-treatment: number analyzed (Participants) | 58 | 49
  Count Variability at Post-treatment | 393.58 (223.01) | 371.08 (310.24)
  Count Mean at 6-month follow-up: number analyzed (Participants) | 57 | 53
  Count Mean at 6-month follow-up | 1362.37 (598.01) | 1281.35 (667.83)
  Count Variability at 6-month follow-up: number analyzed (Participants) | 57 | 53
  Count Variability at 6-month follow-up | 447.2 (257.81) | 354.96 (212.71)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Waking activity count mean (min): Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.34, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -76.85
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Waking activity count mean (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.28, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -87.15
Statistical Analysis 3: Comparison: UC-DT vs TranS-C; Waking activity count variability (min) : Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.18, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.15
Statistical Analysis 4: Comparison: UC-DT vs TranS-C; Waking activity count variability (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.02, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.27

11. Secondary Outcome: Impairment (World Health Organization Disability Assessment Schedule 2.0)
Description: World Health Organization Disability Assessment Schedule 2.0 (WHODAS-2.0). 36-item measure that assesses disability in adults ages 18 years and older. It assesses disability across six domains on a scale from 1-5 (none to extreme or cannot do). Each item on the self-administered version of the WHODAS-2.0 asks the individual to rate how much difficulty he or she has had in specific areas of functioning during the past 30 days. Scores are summed across the six domains (cognition, mobility, self-care, getting along, life activities, and participation). Total scores range from 36 to 180, with higher scores indicating greater levels of disability.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
score on a scale
  Pre-treatment | 81.53 (25.56) | 76.48 (21.38)
  Post-treatment: number analyzed (Participants) | 58 | 49
  Post-treatment | 81.48 (26.80) | 68.93 (25.53)
  6-month follow-up: number analyzed (Participants) | 57 | 53
  6-month follow-up | 73.45 (26.14) | 66.63 (23.17)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.09, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -7.19
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.79, Intent-to-treat, multilevel modeling; Using intent-to-treat, multilevel modeling with maximum likelihood estimation with the assumption of missing at random, to examine continuous outcome; Time by treatment interaction coeff. = -1.13

12. Secondary Outcome: Overall Health ('Healthy Days' Core Module)
Description: Four question 'healthy days' core module developed by the Centers for Disease Control and Prevention. A summary measure combines physically and mentally unhealthy days. An "unhealthy days" summary measure based on the second and third questions and estimates the overall number of recent days (in the past 30 days) when physical or mental health was not good.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
Days
  Pre-treatment | 3.57 (1.17) | 3.44 (1.03)
  Post-treatment: number analyzed (Participants) | 58 | 49
  Post-treatment | 3.40 (1.26) | 3.37 (1.27)
  6-month follow-up: number analyzed (Participants) | 57 | 53
  6-month follow-up | 3.40 (1.26) | 3.37 (1.27)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.46, Intent-to-treat, multilevel modeling; Using intent-to-treat, multilevel modeling with maximum likelihood estimation with the assumption of missing at random, to examine continuous outcome,; Time by treatment interaction coeff. = 0.16
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.10, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.34

13. Secondary Outcome: Composite Sleep Health Score
Description: Composite Sleep Health Score is defined as the sum of scores on 6 sleep health dimensions: Regularity (Midpoint sleep fluctuation across a 7-day sleep diary < 1 hour), Satisfaction (Sleep quality question on PROMIS-Sleep Disturbance (PROMIS = Patient-Reported Outcomes Measurement Information System)), Alertness (Daytime sleepiness question on PROMIS-Sleep Related Impairment (PROMIS = Patient-Reported Outcomes Measurement Information System)), Timing (Mean midpoint sleep across the 7 day sleep diary between 2 and 4 AM), Efficiency (Average sleep efficiency based on the 7 day sleep diary ≥ 85%), and Duration (Total Sleep Time average based on 7 day sleep diary between 7 and 9 hours).
  Each dimension was dichotomized such that 1 = good /yes; 0 = poor/no). Total composite sleep health score ranges from 0 to 6, with larger values indicating better sleep health.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
Score on a scale
  Pre-treatment | 2.28 (1.29) | 2.54 (1.60)
  Post-treatment: number analyzed (Participants) | 58 | 49
  Post-treatment | 2.34 (1.33) | 3.45 (1.39)
  6-month follow-up: number analyzed (Participants) | 57 | 53
  6-month follow-up | 2.53 (1.39) | 3.38 (1.64)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.002, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = 0.91
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.03, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = 0.64

14. Secondary Outcome: Means and Variability of Total Sleep Time (Daily Sleep Diary)
Description: Total sleep time (TST), measured as the total amount of sleep obtained by the participant, was reported via sleep diary over 7 consecutive days. Each participant's mean and within-person SD of TST were calculated to assess typical sleep duration and night-to-night variability. Group-level outcomes reflect the average of these participant-level means and SDs.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
Minutes
  TST mean at Pre-treatment | 452.42 (101.37) | 431.06 (111.47)
  TST variability at Pre-treatment | 109.59 (55.14) | 103.96 (46.37)
  TST mean at Post-treatment: number analyzed (Participants) | 58 | 49
  TST mean at Post-treatment | 459.09 (100.16) | 450.71 (92.77)
  TST variability at Post-treatment: number analyzed (Participants) | 58 | 49
  TST variability at Post-treatment | 123.59 (79.11) | 96.50 (97.84)
  TST mean at 6-month follow-up: number analyzed (Participants) | 57 | 53
  TST mean at 6-month follow-up | 465.23 (115.13) | 464.90 (106.54)
  TST variability at 6-month follow-up: number analyzed (Participants) | 57 | 53
  TST variability at 6-month follow-up | 99.30 (52.38) | 90.87 (58.77)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Means of Total sleep time: Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.23, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = 24.85
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; Means of total sleep time: Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.09, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = 34.31
Statistical Analysis 3: Comparison: UC-DT vs TranS-C; Variability of Total sleep time: Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.19, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -19.90
Statistical Analysis 4: Comparison: UC-DT vs TranS-C; Variability of Total sleep time: Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.91, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -1.76

15. Secondary Outcome: Means and Variability of Total Wake Time (Daily Sleep Diary)
Description: Total wake time (TWT), measured as minutes of wakefulness within a sleep period, was reported via sleep diary over 7 consecutive days. Each participant's mean and within-person SD of their TWT were calculated across days to assess means and night-to-night variability. Group-level outcomes reflect the average of these participant-level means and SDs.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
Minutes
  TWT mean at Pre-treatment | 131.89 (80.47) | 124.84 (75.03)
  TWT variability at Pre-treatment | 77.85 (54.92) | 74.04 (46.48)
  TWT mean at Post-treatment: number analyzed (Participants) | 58 | 49
  TWT mean at Post-treatment | 131.29 (116.57) | 84.37 (49.45)
  (TWT variability at Post-treatment: number analyzed (Participants) | 58 | 49
  (TWT variability at Post-treatment | 82.07 (77.64) | 61.33 (62.27)
  TWT mean at 6-month follow-up: number analyzed (Participants) | 57 | 53
  TWT mean at 6-month follow-up | 118.92 (77.55) | 83.55 (65.53)
  TWT variability at 6-month follow-up: number analyzed (Participants) | 57 | 53
  TWT variability at 6-month follow-up | 73.27 (47.70) | 52.69 (52.56)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; TWT mean (min): Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.04, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -39.33
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; TWT mean (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.13, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -28.56
Statistical Analysis 3: Comparison: UC-DT vs TranS-C; TWT variability (min) : Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.21, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -17.57
Statistical Analysis 4: Comparison: UC-DT vs TranS-C; TWT variability (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.25, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -16.05

16. Secondary Outcome: Means and Variability of Bedtime (Daily Sleep Diary)
Description: Bedtime was reported via a 7-day daily sleep diary using a 24-hour decimal format, where times after midnight are expressed as numbers above 24 (ex. 1:30 am is 25.50). Each participant's mean and within-person SD of bedtime across 7 days were computed to capture average bedtime and variability. Group-level outcomes reflect the average of these participant-level means and SDs.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
hours
  Bedtime mean at Pre-treatment | 22.20 (1.95) | 22.17 (2.36)
  Bedtime variability at Pre-treatment | 1.39 (1.06) | 1.28 (0.79)
  (Bedtime mean at Post-treatment: number analyzed (Participants) | 58 | 49
  (Bedtime mean at Post-treatment | 22.39 (1.56) | 22.00 (1.65)
  Bedtime variability at Post-treatment: number analyzed (Participants) | 58 | 49
  Bedtime variability at Post-treatment | 1.41 (1.07) | 1.01 (0.93)
  Bedtime mean at 6-month follow-up: number analyzed (Participants) | 57 | 53
  Bedtime mean at 6-month follow-up | 22.41 (1.88) | 21.96 (2.13)
  Bedtime variability at 6-month follow-up: number analyzed (Participants) | 57 | 53
  Bedtime variability at 6-month follow-up | 1.55 (1.32) | 1.00 (0.68)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; Bedtime (BT) mean: Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.10, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.55
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; BT mean: Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.04, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.71
Statistical Analysis 3: Comparison: UC-DT vs TranS-C; BT variability: Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.20, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.31
Statistical Analysis 4: Comparison: UC-DT vs TranS-C; BT variability: Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.07, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.45

17. Secondary Outcome: Means and Variability of Wake Time (Daily Sleep Diary)
Description: Wake times, using a 24-hour decimal format, were reported daily across 7 days. The mean and within-person SD were calculated for each participant's wake time across days. Group-level outcomes reflect the average of these participant-level means and SDs.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
hours
  Wake time mean at Pre-treatment | 7.90 (1.83) | 7.31 (2.02)
  Wake time variability at Pre-treatment | 1.42 (0.88) | 1.34 (1.00)
  Wake time mean at Post-treatment: number analyzed (Participants) | 58 | 49
  Wake time mean at Post-treatment | 8.26 (2.25) | 7.31 (1.82)
  Wake time variability at Post-treatment: number analyzed (Participants) | 58 | 49
  Wake time variability at Post-treatment | 1.61 (1.11) | 1.10 (1.08)
  Wake time mean at 6-month follow-up: number analyzed (Participants) | 57 | 53
  Wake time mean at 6-month follow-up | 7.95 (1.83) | 7.33 (1.74)
  Wake time variability at 6-month follow-up: number analyzed (Participants) | 57 | 53
  Wake time variability at 6-month follow-up | 1.22 (0.69) | 1.26 (0.95)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; WT mean: Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.39, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.33
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; WT mean: Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.96, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.02
Statistical Analysis 3: Comparison: UC-DT vs TranS-C; WT variability: Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.047, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.39
Statistical Analysis 4: Comparison: UC-DT vs TranS-C; WT variability: Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.30, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = 0.20

18. Secondary Outcome: Actigraphy Measured Sleep (TWT)
Description: Actigraphy-derived total wake time (TWT), measured as minutes of wakefulness within a sleep period, was collected daily over a 1-week period. Each participant's mean and within-person SD were calculated across the 7 days. Group-level outcomes reflect the average of these participant-level means and SDs.
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | UC-DT | TranS-C
Number analyzed (Participants) | 60 | 61
Minutes
  TWT mean at Pre-treatment | 91.06 (41.52) | 94.95 (55.18)
  TWT variability at Pre-treatment | 55.65 (51.16) | 54.46 (48.26)
  TWT mean at Post-treatment: number analyzed (Participants) | 58 | 49
  TWT mean at Post-treatment | 91.39 (48.65) | 90.80 (44.85)
  TWT variability at Post-treatment: number analyzed (Participants) | 58 | 49
  TWT variability at Post-treatment | 60.36 (68.61) | 51.72 (41.86)
  TWT mean at 6-month follow-up: number analyzed (Participants) | 57 | 53
  TWT mean at 6-month follow-up | 92.73 (41.87) | 84.51 (45.84)
  TWT variability at 6-month follow-up: number analyzed (Participants) | 57 | 53
  TWT variability at 6-month follow-up | 56.22 (48.70) | 41.41 (30.65)
Statistical Analysis 1: Comparison: UC-DT vs TranS-C; TWT mean (min): Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.66, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -4.42
Statistical Analysis 2: Comparison: UC-DT vs TranS-C; TWT mean (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.19, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -13.34
Statistical Analysis 3: Comparison: UC-DT vs TranS-C; TWT variability (min): Treatment effect on change from pre to post, which is 9-14 weeks after the beginning of treatment; Test type: Superiority; p = 0.77, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.05
Statistical Analysis 4: Comparison: UC-DT vs TranS-C; TWT variability (min): Treatment effect on change from pre to 6-month follow-up; Test type: Superiority; p = 0.20, Intent-to-treat, multilevel modeling; [statistical method as in outcome 1, analysis 1]; Time by treatment interaction coeff. = -0.22

19. Other Pre Specified Outcome: Diagnosis of Psychiatric Disorders (MINI International Neuropsychiatric Interview )
Time Frame: Documenting diagnosis at baseline, 10-14 weeks after the beginning of treatment, and 6-month follow-up, no change predicted
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Diagnosis of Sleep Disorders (Duke Structured Interview for Sleep Disorder, DSM-V)
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Sleep and Circadian Problems Interview
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Insomnia Severity Index
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Hypersomnia Severity Index
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Therapy Process Measure
Description: Credibility Expectancy Questionnaire
Time Frame: Administered at the end of Session 2 of treatment
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Medication and Other Treatment Tracking Form
Time Frame: Stability in baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month followup
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Additional Screen for Sleep Apnea
Description: Snoring, tiredness/sleepiness, observed apneas, hypertension, BMI > 35 kg/m2, age > 50 years, neck circumference > 40 cm, and male gender (STOP-BANG) Questionnaire. 8-item screen for obstructive sleep apnea.
Time Frame: Baseline Only
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Brief Pain Inventory (Short Form)
Description: Current symptoms of chronic pain
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month follow-up
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Clinic Staff Qualitative Assessment
Description: Explore barriers and facilitators to implementing an evidence-based sleep treatment in a community setting
Time Frame: One time at the convenience of clinic staff
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Client Behavior Change Interview
Description: Exploration of barriers and facilitators to behavior change
Time Frame: One time following the completion of the first post-treatment assessment
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Salivary Cytokine Assay
Description: Measure of cytokines present in saliva (e.g., Interleukin (IL) -1 beta, IL-6, IL-8, Tumor necrosis factor (TNF) alpha, and/or C-reactive protein (CRP)) to assess immune function
Time Frame: Change from baseline to post treatment, which is 9-14 weeks after the beginning of treatment, and to 6-month follow-up
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Credibility Evaluation Questionnaire (CEQ)
Description: Client evaluation of treatment
Time Frame: Session 2 and Post treatment, which is 9-14 weeks after the beginning of treatment.
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Patient Recall Task
Description: Participant recall of sleep coaching treatment
Time Frame: Post treatment, which is 9-14 weeks after the beginning of treatment, and 6-month follow-up
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Patient Learning Task (Application and Thoughts Subsections)
Description: Client feedback and application of treatment
Time Frame: Post treatment, which is 9-14 weeks after the beginning of treatment, and at 6-month follow-up
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Useful and Utilized Questionnaire
Description: Measure of sleep coaching elements used/useful to clients
Time Frame: Post treatment, which is 9-14 weeks after the beginning of treatment, and at 6-month follow-up
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Treatment Adherence Rating Scale-Therapist Version
Description: Therapist evaluation of client adherence to treatment
Time Frame: After each treatment session filled out by therapist (8 times)
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Body Weight
Description: To calculate BMI
Time Frame: Pre-treatment, post treatment, which is 9-14 weeks after the beginning of treatment, and at 6-month follow-up
Reporting Status: Not Posted

37. Other Pre Specified Outcome: Height
Description: To calculate BMI
Time Frame: Pre-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months.
Description: All-cause mortality, Serious, and Other Adverse Events were monitored through occasional assessment and self-report.
  All-cause mortality did not occur during treatment in either intervention arm, and events were analyzed separately for each intervention arm. In the TranS-C arm, all-cause mortality occurred before the participant received the allocated treatment. In Usual Care, all-cause mortality occurred after the completion of the post-treatment assessment, but before the 6-month follow-up.
Arm/Group | TranS-C | UC-DT
All-Cause Mortality (participants affected / at risk) | 1/61 | 1/60
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 0/61 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02469233/Prot_SAP_000.pdf